CLINICAL TRIAL: NCT01747941
Title: A Double Blind (3rd Party Open) Randomized, Placebo Controlled, Crossover Dose Escalation Study to Investigate the Safety, Tolerability, Pharmacokinetics of PF-06305591 in Healthy Male and Female Subjects
Brief Title: Study to Investigate the Safety, Tolerability, Pharmacokinetics of PF-06305591 in Healthy Male and Female Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: B5281001
Record Dates: First submitted 2012-12-05; First posted 2012-12-12 (Estimated); Last update posted 2013-05-23 (Estimated); Status verified 2013-05

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Cohort 1 (Experimental): Single ascending oral doses in fasted conditions
  Interventions: Drug: PF-06305591; Drug: Placebo
- Cohort 2 (Experimental): Single ascending oral doses in fasted conditions
  Interventions: Drug: PF-06305591; Drug: Placebo
- Cohort 3 (Experimental): Single ascending oral doses in fed conditions
  Interventions: Drug: PF-06305591; Drug: Placebo

INTERVENTIONS:
Drug: PF-06305591 — single dose, solution
  Arms: Cohort 1
Drug: Placebo — matching placebo
  Arms: Cohort 1
Drug: PF-06305591 — single dose, solution
  Arms: Cohort 2
Drug: Placebo — matching placebo
  Arms: Cohort 2
Drug: PF-06305591 — single dose, solution
  Arms: Cohort 3
Drug: Placebo — matching placebo
  Arms: Cohort 3

SUMMARY:
The study is designed to test safety tolerability and PK of single oral ascending doses of PF-06305591,

ELIGIBILITY:
Inclusion Criteria:

* healthy young subjects
* aged 18-55

Exclusion Criteria:

* Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurologic, or allergic disease (including drug allergies, but excluding untreated, asymptomatic, seasonal allergies at the time of dosing).
* Pregnant or nursing females; females of childbearing potential.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2012-11; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs) | 72 hr

SECONDARY OUTCOMES:
Area Under the Curve From Time Zero to Extrapolated Infinite Time [AUC (0 - 8)] | 72 hr

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, Brussels, Belgium

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B5281001&StudyName=Study%20to%20Investigate%20the%20Safety%2C%20Tolerability%2C%20Pharmacokinetics%20of%20PF-06305591%20in%20Healthy%20Male%20and%20Female%20Subjects%20